CLINICAL TRIAL: NCT07317141
Title: Effectiveness of Early Immunization With Nirsevimab on Preschool Wheezing in France
Brief Title: The Effectiveness of Early Immunisation With Nirsevimab on Preschool Wheezing in France, Based on an Analysis of Data From the French Health System Database.
Acronym: INSPIRATION
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0734
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Infant Wheeze; Preschool Age Children; Asthma Childhood
Keywords: nirsevimab; wheezing disease; infants; preschoolers
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Exposed group of children: all children born between 06/02/2023 and 31/01/2024 and who had received nirsevimab before 6 or 12 months of age depending on the outcomes that will be studied.
  Interventions: Other: Effectiveness of passive immunization with nirsevimab
- Non-exposed: Unexposed group of children: all children born between June 06/02/2023 and 31/01/2024 and who did not received nirsevimab.
  The following matching features will be used to ensure comparability between the two groups: sex, month of birth, department of birth.
  Immunized and non-immunized infants will be matched at a 1:2 ratio.

INTERVENTIONS:
Other: Effectiveness of passive immunization with nirsevimab — The investigators will assess the effectiveness of passive immunization with nirsevimab on the occurrence of wheezing during the preschool period.
  Assessment will be separated in two period of time Infants immunized before 6 Months of age will be assessed for hospitalization for wheezing before 2 years of age Infants immunized before 12 months of age will be assessed for recurrent wheezing before 6 years of age.
  An interim analysis at 4 years of age will be done.
  Groups: Exposed

SUMMARY:
Early respiratory syncytial virus (RSV) bronchiolitis is a well-known contributing factor of mid- and long-term respiratory sequelae in children such as recurrent lower tract respiratory infections (LRTIs), preschool wheezing (PW) or decreased lung function at older ages.

Nirsevimab, a monoclonal antibody against RSV with enhanced neutralizing activity and a prolonged half-life, has shown great potential in reducing short term outcomes such as hospitalization for RSV associated bronchiolitis (estimated adjusted effectiveness against hospitalization to 83.0% (95%CI: 73.4 to 89.2). Other countries that have been using nirsevimab almost exhaustively have reported similar results such as in Galicia.

However, prevention of RSV LRTI or delay RSV infection early in life has not been investigated on respiratory manifestations such early wheezing in infancy (ie before 2 years of age) and recurrent wheezing in preschool period (ie between 2 and 6 years old).

Some recent data have shown that nirsevimab was associated with a reduction of wheezing in the year following its administration (HR: 0.73; 95% CI, 0.58-0.93). Other data have shown that not being infected by RSV during the infancy was associated with 26% lower risk of 5-year current asthma than being infected (5) giving good rational for preventive strategies against RSV to impact midterm respiratory outcomes such as PW and then asthma.

Ongoing observational cohort studies will help investigate the question of mid-term effects, but they will come with a high costs and risk of attrition. Administrative national health claims database could prove to be useful and complementary by studying these types of real world outcomes across lives of children that have been immunized by nirsevimab as shown recently.

Therefore, the investigators aim to study the impact of early nirsevimab administration on wheezing manifestations occurring in infancy and beyond during the preschool years.

Our primary objective is to see if nirsevimab administration during the first six months of life has an impact on hospitalization for wheezing episodes during the second year of life, based on the hypothesis that infants who had received nirsevimab have reduced hospitalization for wheezing during their second year of infancy.

ELIGIBILITY:
Inclusion Criteria:

* - Exposed group of children: all children born between 06/02/2023 and 31/01/2024 and who had received nirsevimab before 6 or 12 months of age depending on the outcomes that will be studied.
* Unexposed group of children: all children born between 06/02/2023 and 31/01/2024 and who did not receive nirsevimab

Exclusion Criteria:

* - Infants born in Overseas Departments and Territories (Guadeloupe, Martinique, Guyana, La Réunion, Mayotte, Saint-Pierre-et-Miquelon, French Polynesia, Nouvelle-Calédonie, Wallis-et-Futuna, French Southern and Antarctic Lands, Clipperton island)
* Same-sex twins, as they cannot be differentiated in the French Medicalization of Information Systems Program (PMSI)
* Infants born between 06/02/2023 and 31/01/2024 in a maternity unit that has not reported data on the immunization with nirsevimab
* Infants whose mother had been vaccinated against RSV during pregnancy
* Infants who received palivizumab immunization
* Date of nirsevimab immunization not provided
* Infants hospitalized for wheezing or RSV+ lower respiratory tract infection before receiving nirsevimab
* Infants who were immunized after 12 months of age for outcomes collected between 2 and 6 years old
* Infants who were immunized after 6 months of age for outcomes collected during the second year of life

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study cohorts will combine individual data from the National Health Data System (SNDS), covering the entire French population, and hospitalization data from the French Medicalization of Information Systems Program (PMSI). The SNDS includes socio-demographic data, outpatient reimbursements (including prescriptions), and inpatient care with diagnoses and procedures. The PMSI provides details on hospital stays, diagnoses, and procedures. All data are linked via unique anonymous identifiers. With an average of 60,000 births per month and a 20% exclusion rate, investigators estimate 576,000 eligible patients, exceeding the required sample size (218,000: 70,000 exposed, 148,000 non-exposed).
Sampling Method: Non-Probability Sample
Enrollment: 218000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for wheezing episodes among infants immunized with nirsevimab (exposed group) vs non-immunized (non-exposed group) | During the second year of life (exactly between 6 and 24 months of age)
  The investigators will compare rates of hospitalization between the two groups. Our primary outcome will be captured by using the asthma-related ICD10 codes J45, J46; bronchiolitis related ICD-10 code J21, respiratory failure J96 and wheezing associated respiratory ill

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided